CLINICAL TRIAL: NCT02164955
Title: A Non-interventional Post Authorisation Registry of Patients Treated With Pomalidomide for Relapsed and Refractory Multiple Myeloma Who Have Received at Least Two Prior Treatment Regimens, Including Both Lenalidomide and Bortezomib, and Have Demonstrated Disease Progression on the Last Therapy
Brief Title: A Post Authorisation Registry of IMNOVID (Pomalidomide) for Patients With Relapsed and Refractory Multiple Myeloma.
Status: Completed | Type: Observational
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: CC-4047-MM-015
Record Dates: First submitted 2014-06-13; First posted 2014-06-17 (Estimated); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Multiple Myeloma
Keywords: Pomalidomide; Multiple Myeloma; Relapsed, Refractory; Observational; Imnovid; Registry; Post-approval; Safety
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — pomalidomide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Relapsed and Refractory Multiple Myeloma Patients: Single Cohort of Relapsed and Refractory Multiple Myeloma Patients treated with IMNOVID (pomalidomide)
  Interventions: Drug: IMNOVID

INTERVENTIONS:
Drug: IMNOVID — IMNOVID (pomalidomide) as prescribed in routine clinical practice
  Other Names: pomalidomide; CC-4047; BMS-986379

SUMMARY:
This registry is a prospective, multi-center, observational study and will collect safety data on multiple myeloma adult patients who have received at least two prior therapies and take IMNOVID (pomalidomide) as part of standard care.

The registry will remain open until 500 patients will have received at least 3 cycles of pomalidomide. All patients registered will be followed for up to 3 years after the informed consent date or until death or withdrawal of consent. During this time the incidence of second primary malignancies (SPM), overall survival and any occurrence of a pregnancy will be assessed.

ELIGIBILITY:
Inclusion Criteria:

Understand and voluntarily sign an informed consent form, if applicable, and have never been previously treated with pomalidomide before their inclusion in the Registry.

Patients with symptomatic, measurable relapsed and refractory multiple myeloma who have received at least two prior treatment regimens, including both bortezomib and lenalidomide and have demonstrated disease progression on the last therapy and are commencing a pomalidomide based treatment.

Exclusion Criteria:

Refusal to participate in the Registry or currently participating in the treatment phase of an interventional clinical trial.

Pregnancy.

Women of childbearing potential, unless all the conditions of the pregnancy prevention program are met.

Male patients unable to follow or comply with the required contraceptive measures.

Hypersensitivity to the active substance or to any of the excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic, measurable relapsed and refractory multiple myeloma who have received at least two prior treatment regimens, including both bortezomib and lenalidomide and have demonstrated disease progression on the last therapy and are commencing a pomalidomide based treatment.
Sampling Method: Non-Probability Sample
Enrollment: 775 (Actual)
Dates: Start 2014-06-26 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Determine incidence of risks as outlined in the Risk Management Plan | Up to 3 years
  To characterize and determine the incidence of important identified and potential risks as outlined in the risk management plan (RMP) among previously treated multiple myeloma patients who are currently being treated with IMNOVID (pomalidomide) in a post-marketing setting.

SECONDARY OUTCOMES:
Pregnancy Prevention Programme Effectiveness | Up to 3 years
  To describe and assess the effectiveness, implementation and compliance of the Celgene Pregnancy Prevention Programme for patients recruited in this registry
Previous Treatments | Approximately 6 months
  To describe the type of myeloma treatment administered immediately prior to receiving IMNOVID (pomalidomide).

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (122):
- Belgium (9):
  - Cliniques Universitaires Saint Luc, Brussels, Avenue Hippocrate 10
  - Ziekenhuis Netwerk Antwerpen- Campus Middelheim, Antwerp, Lindendreef 1
  - Az Nikolaas, Sint-Niklaas, Lodewijk de Meesterstraat 5
  - Centre Hospitalier Peltzer-La Tourelle, Verviers, Rue Du Parc 29
  - Centre hospitalier de Jolimont, La Louvière, Rue Ferrer 159
  - Les Cliniques Du Sud Luxembourg- Clinique Saint-Joseph, Arlon
  - Universitair Ziekenhuis Antwerpen, Edegem
  - CHC, Liège
  - Clinique Saint-Pierre, Ottignies
- Denmark (3):
  - Odense Hospital, Odense, Kloevervanget 10
  - Aarhus Universitetshospital, Karup, Noerrebrogade 44
  - Vejle Hospital, Dep of hema Kabbeltoft, Kabbeltoft 25, Vejle
- Germany (27):
  - Gemeinschaftspraxis Fur Hamatologie Und Onkologie, Koln-Kalk, Buchforststr 14
  - Charite der Humboldt-Universität, Berlin, Chariteplatz 1
  - Klinikum Enroll von Bergmann, Potsdam, Charlotteustr 72
  - Klinikum Traunstein, Traunstein, Cuno-Niggl-Strate 3
  - Studienzentrum Haematologie/Onkologie/Diabetologie, Aschaffenburg, Elisenstr.26
  - Universitaetsklinikum Essen, Westdeutsches Tumorzentrum, Essen, Hufelandstraße 55
  - Diakonie-Klinikum Schwabisch Hall, Schwäbisch Hall, Innere Medizin III
  - UBAG MVZ Mitte/ MVZ Delitzsch GmbH, Delitzsch, Ludwig- Jahn- Str. 4
  - Klinikum Grosshadern-Klinikum Der Ludwig-Maximilian Universitaet Muenchen, München, Marchioninistr. 15
  - Stadtisches Klinikum Karlsruhe, Karlsruhe, Medizinische Klinik III
  - Schwerpunktpraxis und Tagesklinik fur Hamatologie und Onkologie, Kronach, Niederbronner Stabe 2
  - Klinikum Lippe-Lemgo, Minden, Rintelner Strae 85
  - HELIOS Klinikum Berlin-Buch, Berlin, Schwanebecker Chaussee 50
  - Malteser Krankenhaus St. Franziskus Hospital, Flensburg, Waldstr. 17
  - Dr. Reiner Weinberg, Md, Office Of, Aachen, Weberstr. 8
  - Evangelisches Krankenhaus Hamm GgmbH, Hamm, Werler Str. 110
  - Carl-Thiem-Klinikum Cottbus, Cottbus
  - Klinikum Frankfurt Höchst, Klinik für Innere Medizin 3, Frankfurt
  - GP Dres. Verpoort, Hamburg
  - Uberortliche Gemeinschaftspraxis - Schwerpunkt Haematologie, internistische Onkologie & Palliativmedizin, Dres. Verpoort, Wierecky & Zeller, Hamburg
  - Praxis Dr Schwarzer, Leipzig
  - Johannes Wesling Klinikum Minden, Minden
  - Klinik für Hämatologie, Onkologie und Palliativmedizin Mühlenkreiskliniken, Johannes Wesling Klinikum Minden, Minden
  - Gemeinschaftspraxis für, Hämato-Onkologie am St. Josef, Krankenhaus Moers, Moers
  - Stauferklinikum Schwaebisch Gmuend, Mutlangen
  - Zentrum für Innere Medizin, Mutlangen
  - Studienzentrum Onkologie Ravensburg, Ravensburg
- Italy (25):
  - Laboratorio Analisi Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo, FG
  - AOUC Azienda Ospedaliero-Universitaria Careggi, Florence, Florence
  - Reparto Di Ematologia Dell'Azienda, Brescia, Lombardy
  - Azienda Ospedaliera Di Rilievo Nazionale (AORN) 'Antonio Cardarelli', Napoli, Naples
  - Institute of Hematology- Sapienza University -Rome, Italy, Roma, Rome
  - Azienda Ospedaliera Universitaria di Padova, Padua, Veneto
  - Azienda Ospedaliera Univarsitaria Consorziale Policlinico di Bari, Bari
  - Azienda Ospedaliera Ospedali Riuniti di Bergamo, Bergamo
  - AOU-S.Orsola-Malpighi - Universita degli Studi di Bologna, Bologna
  - Azienda Ospedaliera Spedali Civili di Brescia-Universita degli Studi Di Brescia, Brescia
  - Centro Trapianti Midollo Osseo Ospedale Bnaghi, Cagliari
  - A.O.U. Vittorio Emanuele di Catania-Ospedale Ferrarotto, Catania
  - Azienda Ospedaliera Universitaria "San Martino", Genova
  - Ospedale San Raffaele Srl, Milan
  - Ematologia, Policlinico di Milano, Milan
  - Casa di Cura La Maddalena, Palermo
  - AOUP, Santa Chiara Hospital, Pisa
  - A.O. Bianchi Melacrino Morelli, Reggio Calabria
  - Arcispedale S. Maria Nuova, Reggio Emilia
  - Policlinico S.Eugenio, Roma
  - A.O.U.S. Giovanni e Ruggi d'Aragona UOC UTIC, Salerno
  - AOU Ospedali Riuniti Umbertio I, Torrette Di Ancona
  - U.O Ematologia Az. ULSS9 di Treviso, Treviso
  - Unita di Oncologia Polmonare A.o. San, Turin
  - Universita Degli Studi Policlinico, Udine
- Norway (4):
  - HF Alesund Hospital, Ålesund
  - Helse Bergen HF Haukeland University Hospital, Bergen
  - Vestre Viken/Baerums sjukhus, Drammen
  - Fredrikstad Hospital, Fredrikstad
- Spain (22):
  - Hospital Costa Del Sol, Marbella, Autovia A-7, Km 187
  - University Hospital Reina Sofia, Córdoba, Avda Menendez Pidal S/n
  - Nuestra Senora de Valme, Seville, Avda. Bellavista, S/N
  - Hospital Puerta del Mar, Cadiz, Avenida Ana de Viya, 21
  - Hospital Universitario Central de Asturias, Oviedo, Avenida de Roma S/n
  - General de Jane, Jaén, Avenida Ejercito Espanol 10
  - General San Pedro de Alcantara, Cáceres, Avenida Pablo Naranjo Porras
  - Hospital Clinico Universitario De Valladolid, Valladolid, Avenida Ramon Y Cajal 3
  - Hospital Universitario de La Princesa, Madrid, C/ Diego de León 62, 3a Planta
  - Hospital Xeral de Lugo, Lugo, C/ Doctor Severo Ochoa S/N
  - Hospital Son Dureta, Palma de Mallorca, Calle Andrea Doria 55
  - Hospital General Universitario Santa Lucia, Cartagena (murcia), Calle Mezquita
  - Hospital Arnau De Vilanova De Valencia, Valencia, Calle San Clemente, 12
  - Hospital General Universitario de Elche, Elche, CAMI de L´almassera 11
  - Hospital de Cabuenes, Gijón, Camino de Los Prados
  - Hospital Universitario Nuestra Senora De Candelaria, Santa Cruz de Tenerife, Carretera Del Rosario, 145
  - Hospital Fundacion Son Llatzer, Palma de Mallorca, Ctra. Manacor, Km. 4
  - Hospital universitario de Alava, Alava, Jose Achotegui
  - IC0 Duran y Reynalds, Barcelona, L´Hospitalet de Llobregat
  - Hospital Universitari Vall d'Hebron, Barcelona, Passeig de La Vall D'Hebron 119-129
  - Ctra. Orihuela - Almoradi, Orihuela (alicante), S/N San Bartolome
  - Hospital Universitario Virgen de la Victoria, Málaga, Servicio de Oncologia
- Sweden (2):
  - Sunderby Hospital, Luleå
  - University Hospital UMEA, Umeå
- United Kingdom (30):
  - Pinderfields Hospital-Mid Yorkshire Nhs Trust, Wakefield, Aberford Road
  - Doncaster Royal Infirmary - Doncaster And Bassetlaw Hospitals Nhs Foundation Trust, Doncaster, Armthorpe Road
  - Northhampton Gerneral Hospital, Northampton, Cliftonville
  - County Durham and Darlington NHS foundation Trust, County Durham, Darlington Memorial Hospital
  - Broomfield Hospital, Broomfield,Chelmsford, Essex
  - Aberdeen Royal Infirmary - Nhs Grampian, Aberdeen, Foresterhill Road
  - The Newcastle Upon Tyne Hospitals Nhs Foundation, Newcastle upon Tyne, Freeman Hospital
  - Lincoln County Hospital - United Lincolnshire Hospitals Nhs Trust, Lincoln, Greetwell Road
  - Maidstone Hospital - Maidstone And Tunbridge Wells Nhs Trust-Kent Oncology Centre, Maidstone, Kent
  - Blackpool Victoria Hospital - Blackpool, Fylde And Wyre Hospitals Nhs Foundation Trust, Blackpool, Lancashire
  - Huddersfield Royal Infirmary - Calderdale And Huddersfield Nhs Foundation Trust, Huddersfield, Lindley
  - Worthing Hospital - Western Sussex Hospitals Nhs Trust, Worthing, Lyndhurst Road
  - Monklands Hospital Trust: Nhs Lanarkshire - Acute Services Division, Airdrie, Monkscourt Avenue
  - Southmead Hospital - North Bristol Nhs Trust Recruiting, Bristol, Southmead Road
  - City Hospitals Sunderland NHS Trust Recruiting, Sunderland, Sunderland Royal Hospital
  - Colchester General Hospital - Colchester Hospital University Nhs Foundation Trust, Colchester, Turner Road
  - University Hospital of Wales, Cardiff, Vale Of Glamorgan
  - Northwick Park Hospital - North West London Hospitals Nhs Trust, Harrow, Watford Road
  - Singleton Hospital - Abertawe Bro Morgannwg University Nhs Trust, Swansea, West Glamorgan
  - Worcestershire Acute Hospitals NHS Trust - Worcestershire Royal Hospital, Worcester, Worcestershire
  - St Helier Hospital - Epsom and St Helier University Hospitals NHS Trust, Carshalton, Wrythe Lane
  - Basingstoke and North Hampshire Hospital, Basingstoke
  - Royal United Hospital, Bath - Royal United Hospital Bath NHS Trust, Bath
  - Dorset County Hospital, Dorchester
  - The Royal Liverpool and Broadgreen -University Hospitals NHS, Liverpool
  - Specialist Cancer Pharmacist-Oxford Cancer Centre & Cancer Research UK-Churchill Hospital-Oxford University Hospitals NHS Trust, Oxford
  - Royal Berkshire hospital, Reading
  - Wexham Park Hospital, Slough
  - Royal Cornwall Hospital, Truro
  - Northumbria Healthcare NHS Foundation Trust North Tyneside Hospital, Tyne and Wear

REFERENCES:
- [Background] Moreau P, Dimopoulos MA, Richardson PG, Siegel DS, Cavo M, Corradini P, Weisel K, Delforge M, O'Gorman P, Song K, Chen C, Bahlis N, Oriol A, Hansson M, Kaiser M, Anttila P, Raymakers R, Joao C, Cook G, Sternas L, Biyukov T, Slaughter A, Hong K, Herring J, Yu X, Zaki M, San-Miguel J. Adverse event management in patients with relapsed and refractory multiple myeloma taking pomalidomide plus low-dose dexamethasone: A pooled analysis. Eur J Haematol. 2017 Sep;99(3):199-206. doi: 10.1111/ejh.12903. Epub 2017 Jun 14. PMID 28504846
- [Background] Schafer PH, Ye Y, Wu L, Kosek J, Ringheim G, Yang Z, Liu L, Thomas M, Palmisano M, Chopra R. Cereblon modulator iberdomide induces degradation of the transcription factors Ikaros and Aiolos: immunomodulation in healthy volunteers and relevance to systemic lupus erythematosus. Ann Rheum Dis. 2018 Oct;77(10):1516-1523. doi: 10.1136/annrheumdis-2017-212916. Epub 2018 Jun 26. PMID 29945920
- [Background] Dinner S, Dunn TJ, Price E, Coutre SE, Gotlib J, Berube C, Kaufman GP, Medeiros BC, Liedtke M. A phase I, open-label, dose-escalation study of amrubicin in combination with lenalidomide and weekly dexamethasone in previously treated adults with relapsed or refractory multiple myeloma. Int J Hematol. 2018 Sep;108(3):267-273. doi: 10.1007/s12185-018-2468-5. Epub 2018 May 25. PMID 29802551
- See also: Expanded Access for CC-4047 — https://clinicaltrials.gov/ct2/show/NCT03723096?term=NCT03723096&rank=1